CLINICAL TRIAL: NCT00295802
Title: Ablatherm Integrated Imaging High Intensity Focused Ultrasound for the Indication of Low Risk, Localized Prostate Cancer
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: EDAP TMS S.A. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: G050103
Record Dates: First submitted 2006-02-22; First posted 2006-02-24 (Estimated); Last update posted 2014-02-07 (Estimated); Status verified 2014-02

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; HIFU; EDAP; Low Risk, Localized Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Cryotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- HIFU (Experimental): Integrated Imaging High Intensity Focused Ultrasound using the Ablatherm Device
  Interventions: Device: Integrated Imaging High Intensity Focused Ultrasound
- Cryotherapy (Active Comparator): Endocare CRYOcare Cryosurgical and Galil Medical CRYO-HIT Systems (cryotherapy)
  Interventions: Device: Endocare CRYOcare Cryosurgical and Galil Medical CRYO-HIT Systems (cryotherapy)

INTERVENTIONS:
Device: Integrated Imaging High Intensity Focused Ultrasound
  Other Names: HIFU
  Arms: HIFU
Device: Endocare CRYOcare Cryosurgical and Galil Medical CRYO-HIT Systems (cryotherapy) — Cryotherapy
  Other Names: Endocare CRYOcare Cryosurgical; Galil Medical CRYO-HIT Systems (cryotherapy)
  Arms: Cryotherapy

SUMMARY:
The purpose of this study is to determine the substantial equivalence of the Ablatherm high intensity focused ultrasound (HIFU) as compared to cryotherapy for the treatment of low risk, localized prostate cancer.

DETAILED DESCRIPTION:
Primary hypothesis of this clinical investigation is that HIFU with the Ablatherm Integrated Imaging is non-inferior to minimally invasive cryosurgery as an effective treatment method for low risk, localized prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of prostate cancer confirmed by PSA and prostate biopsy
* Male subjects, aged equal to or over 50 years
* Organ-confined prostate cancer, clinical stage T1a, b, or c or T2a
* At least one positive biopsy within the previous 6 months
* PSA equal to or less than 10 ng/ml
* Gleason score equal to or less than 6
* Histological grading of 3+3, 3+2, 2+3, 2+4, or 2+2 based upon the baseline transrectal ultrasound (TRUS)-guided 10 core biopsy results. A subject with a histological grading of primary 4 will not be permitted for study enrollment.
* Prostate volume equal to or less than 40 cc
* Prostate anteroposterior (AP) diameter equal to or less than 25 mm
* Normal rectal anatomy and rectal mucosa
* Maximum rectal wall measurement 6 mm
* The Investigator has completed a medical history and a physical examination to assure that the subjects meet all study enrollment criteria
* The subject is willing and able to read, understand, and sign the study specific informed consent form
* The subject agrees to comply with study protocol requirements, including HIFU or cryotherapy treatment and all follow up visit requirements through 24 months of follow up treatment.

Exclusion Criteria:

* Evidence of seminal vesicle involvement
* Evidence of lymph node involvement or metastasis
* Any previous treatment for prostate cancer including: external beam radiation therapy (EBRT), hormone therapy and/or previous bilateral orchiectomy
* Previous surgery or procedure of the prostate (except prostate biopsy) or urethra within the prior one year
* Calcification inducing a shadow in the prostate which cannot be included in the targeted volume
* Large median lobe of the prostate which cannot be included in the target volume
* Use within the previous 2 months of finasteride
* Previous rectal surgery (other than hemorrhoidectomy) or history of rectal disease
* Active inflammatory bowel syndrome
* Current superficial bladder cancer, urethral stricture, or bladder neck contracture
* Active urinary tract infection or prostatitis (the subject may be enrolled once the infection has been treated and has resolved)
* Compromised renal function or upper urinary tract disease as a result of urinary obstruction
* A history of bleeding disorders/coagulopathy or ongoing treatment for this condition
* Urinary tract or rectal fistula
* Rectal fibrosis, rectal stenosis, or other anomalies making the Ablatherm Integrated Imaging rectal probe insertion difficult
* Anatomical anomaly of the rectum or anomaly of the rectal mucous membrane
* Prostate seroma, prostate abscess, or urethral stenosis
* An intraprostatic implant such as a stent or catheter, or any implant or prosthesis at less than 1 cm from the prostate
* Interest in future fertility
* Concurrent illness, disability, or geographical residence would hamper attendance at required study visits
* Known latex hypersensitivity
* Current participation in another clinical investigation of a medical device or a drug or has participated in such a study within 30 days prior to study enrollment
* The Investigator believes that the subject will be unwilling or unable to comply with study protocol requirements, including the HIFU or cryotherapy procedure and study-related follow up visit requirements.

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2006-04; Primary Completion 2012-08 (Actual); Study Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
Attainment achievement of prostate-specific antigen (PSA) nadir < 0.5 ng/ml and stability of PSA according to American Society for Therapeutic Radiology and Oncology (ASTRO) criteria through 24 month follow up without a positive biopsy | Through 24 month period

SECONDARY OUTCOMES:
Achievement of a nadir PSA within 6 months < 0.5 ng/ml | 6 months
Overall survival, defined as time to death due to any cause | From date of treatment until the date of death due to any cause
Disease specific survival, defined as the time to death due to the underlying disease | "From date of treatment until the date of death due to the underlying cause
Change from baseline in the University of California, Los Angeles Quality of Life (UCLA QOL) | 1 month, 6 months, 12 months, 24 months
Change from baseline in the International Prostate Symptom Score (IPSS) | 1 month, 6 months, 12 months, 24 months

OTHER OUTCOMES:
The occurrence of adverse events and device-related adverse events reported | through out study

CONTACTS AND LOCATIONS:
Overall Officials: Carey Robertson, MD, Principal Investigator — Duke University
Locations (15):
- United States (14):
  - Chinn & Chinn Urology Associates, Arcadia, California
  - Univeristy of Colorado Hospital and Health Science Center, Aurora, Colorado
  - Florida Foundation for Healthcare Research Inc, Ocala, Florida
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Brooklyn Urology Research Group, Brooklyn, New York
  - Sloan-Kettering Institute, New York, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Urolgoy Associates of North Texas, Arlington, Texas
  - The University of Texas M.D. Anderson Cancer Center, Houston, Texas
  - Virginia Urology Center, Richmond, Virginia
  - Medical College of Wisconsin, Inc., Milwaukee, Wisconsin
- Maple Leaf HIFU, Hamilton, Ontario, Canada

REFERENCES:
- [Background] Thuroff S, Chaussy C, Vallancien G, Wieland W, Kiel HJ, Le Duc A, Desgrandchamps F, De La Rosette JJ, Gelet A. High-intensity focused ultrasound and localized prostate cancer: efficacy results from the European multicentric study. J Endourol. 2003 Oct;17(8):673-7. doi: 10.1089/089277903322518699. PMID 14622488